CLINICAL TRIAL: NCT07172958
Title: Selective Antigen Specific dTβRII-expressing T Cells and B7-H3 CAR T Cells in Subjects With Relapsed/Refractory Embryonal Tumors (SABRE)
Brief Title: Selective Antigen Specific T Cells and CAR T Cells in Subjects With Relapsed/Refractory Embryonal Tumors (SABRE)
Acronym: SABRE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer Research UK (Other); The Mark Foundation for Cancer Research (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001593
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rhabdomyosarcoma; Ewing Sarcoma; Neuroblastoma; Wilms Tumor
Keywords: CAR T Therapy for Embryonal tumors; T cell Therapy for Embryonal tumors
MeSH Terms: conditions — Rhabdomyosarcoma; Sarcoma, Ewing; Neuroblastoma; Wilms Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- This is single arm study. (Experimental): Lymphodepleting chemotherapy regimen with cyclophosphamide and fludarabine will be administered prior to CAR-TA T cell product infusion. The DNR-TA T cells and B7-H3 CAR T cells will be generated and combined into a final product comprised of the two T cell components combined at a 1:1 ratio.
  Interventions: Biological: Selective Antigen Specific dTβRII-expressing T cells combined with B7-H3 CAR T cells

INTERVENTIONS:
Biological: Selective Antigen Specific dTβRII-expressing T cells combined with B7-H3 CAR T cells — Selective Antigen Specific dTβRII-expressing T cells combined with B7-H3 CAR T cells

SUMMARY:
This is a phase I dose-escalation study to determine the safety and feasibility of autologous CAR-TA T cells (B7-H3 CAR+ T cells administered with DNR-PRAME Tumor Antigen-specific T cells) following lymphodepleting chemotherapy in participants with relapsed/refractory rhabdomyosarcoma, Ewing sarcoma, neuroblastoma and Wilms tumor.

Patients will be enrolled to one of three planned dose levels with B7-H3 CAR T cell dose determined based on the percentage of B7-H3 transduced cells (B7-H3+ population of cells), and dTBRII-transduced PRAME TA-specific T cell dose based on the total cell population. Both doses will be based on the recipient's body weight.

The safety of the CAR-TA T cell product will be evaluated and the maximum tolerated dose (MTD) will be determined. The safety endpoint will be assessed by monitoring for dose limiting toxicities for 28 days following CAR-TA T cell administration.

DETAILED DESCRIPTION:
This protocol is designed as a phase I dose-escalation study. Procurement phase: During the procurement phase of this protocol, upon SABRE Procurement Consent and procurement eligibility confirmation, participants will undergo a non-mobilized apheresis for collection of mononuclear cells to be used for the CAR-TA T cell product manufacturing.

Treatment phase: Once the CAR-TA T cell products are released and patients are confirmed eligible for CAR-TA T cell product infusion, participants will undergo protocol therapy at Children's National Hospital, consisting of a standard Lymphodepleting chemotherapy preparative regimen with fludarabine and cyclophosphamide, followed by intravenous infusion of the combined CAR-TA T cell product. The DNR-TA T cells and B7-H3 CAR T cells will be generated and combined into a final product comprised of the two T cell components combined at a 1:1 ratio. Patients will be enrolled to one of three CAR-TA T cell product dose levels (dose levels 1, 2 and 3). There are provisions in place to dose de-escalate for safety concerns (dose level -1).

Fludarabine will be administered intravenously once daily over 30 minutes, days -5 through -2 (4 doses in total). The dose of fludarabine will be 30 mg/m2 /day. Cyclophosphamide will be administered intravenously once daily over 30 minutes, days -5 and -4 (2 doses in total). The dose of cyclophosphamide will be 500 mg/m2 /day.

The first 3 patients enrolled on study will be ≥ 12 years of age at enrollment and treated at dose level 1 (1 x 10e6/kg). If no DLTs are observed in this cohort, enrollment at dose levels 2 (3 x 10e6/kg) and 3 (10 x 10e6/kg) will expand to include patients aged ≥ 1 year and < 24 years.

Patients will remain admitted for at least 7 days following the CAR-TA T cell infusion. All infused patients will be followed with weekly visits during the 28-day dose-limiting toxicity monitoring period where they will be clinically assessed, and safety and research blood draws will be performed.

Ideally, patients should not receive other systemic or local cancer-directed therapies for at least 28 days after the CAR-TA T cell infusion.

Participants will be followed closely for 1 year following the CAR-TA T-cell infusion. After 1 year, yearly assessments will be done up to 15 years. The visits will consist of labs and examinations as well as talking to participants about how they are feeling. Participants will be followed for toxicity until the last follow-up post CAR-TA T cell product administration.

This study will be conducted at Children's National Hospital (CNH). Cell culture manipulations will be carried out in the CETI Good Manufacturing Practice (GMP) facility within Children's National Hospital using current standard operating procedures (SOPs).

Up to 18 participants will be treated on this protocol to meet the primary objective over an estimated accrual period of 5 years

ELIGIBILITY:
Inclusion Criteria:

Recipient Inclusion Criteria for Procurement:

* Diagnosis of relapsed/refractory rhabdomyosarcoma, Ewing sarcoma, neuroblastoma, or Wilms tumor
* Refractory disease, residual detectable disease or relapsed disease following available standard of care therapies with known clinical benefit for their specific tumor type, or unable to receive such therapies due to unacceptable toxicity or contraindication
* Measurable or evaluable disease by imaging, as determined following most recent therapy
* Age ≥ 1 year and < 24 years
* Weight > 10 kg
* No systemic steroid exposure within 1 week of procurement
* Karnofsky/Lansky score of ≥ 60 (See Appendix 3)
* Participants of childbearing potential or capable of fathering a child must agree to use effective contraceptive measure/s (as described in Appendix 5) during study protocol participation through 6 months following the administration of the CAR-TA T cells
* ANC > 500/µL
* ALC > 1000/µL
* Platelet count > 50,000/uL (level can be achieved with transfusion)
* Bilirubin ≤ 2.5 mg/dL
* Aspartate aminotransferase (AST)/Alanine transaminase (ALT) ≤ 5x the upper limit of normal for age
* Serum creatinine Maximum serum creatinine (mg/dL) Age Male Female

  1. to < 2 years 0.6 0.6
  2. to < 6 years 0.8 0.8

  6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.2

  ≥ 16 years 1.7 1.4 OR Creatinine clearance or glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m for patients with levels above
* For FOCBP: Negative pregnancy test
* Pulse oximetry of > 90% on room air
* Adequate cardiac function defined as: o Shortening fraction of ≥ 27% by echocardiogram, or o Ejection fraction of > 50% by echocardiogram or radionuclide angiogram (i.e., MUGA).
* No acute neurological toxicity > grade 1 (with the exception of peripheral sensory neuropathy or controlled seizure disorder on anti-epileptics).
* The following time frames must have elapsed between prior therapy completion and apheresis cell collection:

  * Myelosuppressive chemotherapy/immunomodulatory medications: At least 3 weeks, or 6 weeks if prior nitrosourea.
  * Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor. At least 14 days after receiving pegfilgrastim.
  * Biological agent, tyrosine kinase inhibitor, targeted agent, metronomic chemotherapy: At least 7 days since the completion of therapy with a biologic agent, tyrosine kinase inhibitor, targeted agent, or metronomic non-myelosuppressive regimen.
  * Monoclonal antibodies and checkpoint inhibitors: At least 3 weeks or 5 half-lives (whichever is shorter) since the last dose of a monoclonal antibody or checkpoint inhibitor.
  * Radiotherapy (XRT): At least 3 weeks since XRT, and at least 6 weeks if radiation involved the CNS or lung fields. Exception: There is no time restriction for palliative radiation with minimal bone marrow involvement and the patient has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression.
  * Autologous stem cell transplant/infusion: At least 6 weeks from their infusion after an autologous stem cell infusion following myeloablative therapy. Patients who received an autologous stem cell infusion following non-myeloablative therapy do not have a wash-out period; they are eligible once they meet all other eligibility requirements, including recovery from acute side effects.
  * Investigational agent: at least 28 days since receiving an investigational agent.
* Patient or parent/guardian capable of providing informed consent.

Recipient Inclusion Criteria for CAR-TA T cell product Infusion:

* No systemic steroid exposure within 1 week prior to protocol therapy initiation
* Karnofsky/Lansky score of ≥ 60 (See Appendix 3)
* ANC > 750/uL
* Platelet count > 75,000/uL
* Bilirubin ≤ 2.5 mg/dL
* AST/ALT ≤ 5x the upper limit of normal for age
* Serum creatinine Maximum serum creatinine (mg/dL) Age Male Female

  1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.2

  ≥ 16 years 1.7 1.4 OR Creatinine clearance or glomerular filtration rate (GFR) ≥ 70 mL/min/1.73 m for patients with levels above
* For FOCBP: Negative pregnancy test
* Participants of childbearing potential or capable of fathering a child must agree to use effective contraceptive measure/s (as described in Appendix 5) through 6 months following the administration of the CAR-TA T cells
* Adequate respiratory function defined as oxygen saturation 90% or higher on room air
* No acute neurological toxicity > grade 1 (with the exception of peripheral sensory neuropathy or controlled seizure disorder on anti-epileptics).
* Adequate cardiac function defined as:

  * Shortening fraction of ≥ 27% by echocardiogram, or
  * Ejection fraction of > 50% by echocardiogram or radionuclide angiogram
* The following time frames must have elapsed between completion of prior therapy and the initiation of SABRE protocol therapy:

  * Myelosuppressive chemotherapy: At least 2 weeks from last dose of chemotherapy.
  * Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor. At least 14 days after receiving pegfilgrastim.
  * Biological agent, tyrosine kinase inhibitor, targeted agent, metronomic chemotherapy: At least 7 days since the completion of therapy with a biologic agent, tyrosine kinase inhibitor, targeted agent, or metronomic non-myelosuppressive regimen.
  * Monoclonal antibodies and checkpoint inhibitors: At least 3 weeks or 5 half-lives (whichever is shorter) since the last dose of a monoclonal antibody or checkpoint inhibitor.
  * Radiotherapy (XRT): At least 3 weeks since XRT, and at least 6 weeks if radiation involved CNS or lung fields. Exception: There is no time restriction for palliative radiation with minimal bone marrow involvement and the patient has measurable/evaluable disease outside the radiation port or the site of radiation has documented progression.
  * Investigational agent: At least 28 days since receiving an investigational agent.
* Patient or parent/guardian capable of providing informed consent.

Exclusion Criteria:

Recipient Procurement Exclusion Criteria:

* Patients with known CNS disease.
* Patients with uncontrolled infection/s or known HIV infection
* Pregnant or lactating females.
* Patients who have undergone previous allogeneic stem cell transplant.

Recipient Exclusion Criteria for CAR-TA T cell product Infusions:

* Patients with uncontrolled infections or known HIV infection.
* Pregnant or lactating females
* Whole lung/mediastinal radiation within 12 weeks
* Clinically significant systemic illness or medical condition likely to interfere with assessment of safety or efficacy

Ages: 1 Year to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Estimated)
Dates: Start 2026-01-27 (Estimated); Primary Completion 2035-12 (Estimated); Study Completion 2038-12 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or more immediate infusion-related adverse event | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 3 or higher immediate infusion-related adverse events, assessed using the Common Terminology Criteria for Adverse Events (CTCAE, version 5.0; Grades 1-5; higher grades indicate worse severity), occurring during or immediately following the CAR-TA T cell infusion.
Grade 4 or more Immune Effector Cell Associated Neurotoxicity Syndrome (ICANS) | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 4 or higher Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS), assessed using the American Society for Transplantation and Cellular Therapy (ASTCT) CRS and ICANS Consensus Grading Criteria (Grades 1-5; higher grades indicate worse severity).
Grade 3 neurotoxicity or ICANS persisting for more than 72 hours | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 3 neurotoxicity or ICANS with a duration greater than 72 hours. (severity grades assessed as per American Society for Transplantation and Cellular Therapy (ASTCT) CRS and ICANS Consensus Criteria)
Grade 4 or more Cytokine Release Syndrome (CRS) | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 4 or higher Cytokine Release Syndrome (CRS), assessed using ASTCT CRS Consensus Grading Criteria (Grades 1-5; higher = worse).
Grade 3 Cytokine Release Syndrome (CRS) lasting more than 14 days | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 3 CRS with a duration greater than 14 days
Grade 3 or more Hemophagocytic Lymphohistiocytosis (HLH) | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 3 or higher Hemophagocytic Lymphohistiocytosis (HLH), assessed using CTCAE v5.0.
Grade 3 or more fever lasting for more than 14 days | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing fever of Grade 3 or higher, persisting longer than 14 days, assessed using CTCAE v5.0.
Grade 4 or more infection uncontrolled for more than 7 days | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing infection of Grade 4 or higher severity that is uncontrolled for more than 7 days, assessed using CTCAE v5.0.
Any unexpected toxicity of Grade 2 or more | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing unexpected toxicities of Grade 2 or higher, assessed using CTCAE v5.0.
Any expected toxicity above Grade 4 | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing expected toxicity above Grade 4 (i.e., Grade 5 toxicity), assessed using CTCAE v5.0.
Any expected toxicity above Grade 3 lasting longer than 72 hours | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing expected toxicity greater than Grade 3, persisting longer than 72 hours, assessed using CTCAE v5.0.
Grade 2 toxicity persisting for more than 7 days AND considered intolerable to the patient and/or not controlled with standard supportive care | Within 28 days from the CAR-TA T cell infusion
  Number of patients experiencing Grade 2 toxicity persisting for more than 7 days that is intolerable to the patient and/or not controlled with standard supportive care, assessed using CTCAE v5.0.

SECONDARY OUTCOMES:
Response to CAR-TA T cell therapy | Up to 5 years from the CAR-TA T cell infusion
  Number of patients who respond to CAR-TA T cell therapy for treatment of relapsed or refractory rhabdomyosarcoma, Ewing sarcoma, neuroblastoma and Wilms tumor, defined as complete response, partial response, or stable disease following infusion of the CAR-TA T cell product. Disease response will be assessed using protocol-specified criteria.
Progression-free survival | Up to 12 months from the CAR-TA T cell infusion
  Time from infusion of the investigational product to the first documented disease progression or death from any cause
Overall survival | Up to 12 months from the CAR-TA T cell infusion
  Time from the from infusion of the investigational product to death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Holly Meany, MD, Principal Investigator — Children's National Research Institute; Amy Hont, MD, Principal Investigator — Children's National Research Institute
Locations (2):
- United States (2):
  - Children's National Hospital, Washington D.C., District of Columbia
  - Childrens National Hospital, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: No